CLINICAL TRIAL: NCT04716673
Title: Investigating the Effect of Closed-loop Auditory Stimulation on Sleep and Behavior in Patients With Epilepsy and Healthy Controls: a Developmental Study
Brief Title: Stimulation of Sleep in Patients With Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: ETH Zurich (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2019-02134
Record Dates: First submitted 2020-12-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Epilepsy
Keywords: epilepsy; sleep; closed-loop auditory stimulation; epileptic discharges; spikes
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: The investigators aim to evaluate the effect of closed-loop auditory stimulation during sleep in healthy children, adolescents and adults, as well children, adolescents and adults with epilepsy. During closed-loop auditory stimulation, a brief, quiet, non-arousing auditory stimuli, e.g. brief bursts of pink noise (50ms), are presented at specific moments during sleep (STIM condition). This procedure allows to noninvasively interact with endogenous brain activity and to influence sleep-dependent neuroplasticity. During one experimental night, closed-loop auditory stimulation will be applied (STIM night). In the SHAM night, the experimental set-up is the same as in the experimental night, but no sounds will be presented.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study helpers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Children (4-11y) with epilepsy (Experimental): Down-phase-targeted closed-loop auditory stimulation is administered in each arm.
  Interventions: Other: Down-phase targeted auditory stimulation
- Teenagers (12-17y) with epilepsy (Experimental)
  Interventions: Other: Down-phase targeted auditory stimulation
- Young adults (18-30y) with epilepsy (Experimental)
  Interventions: Other: Down-phase targeted auditory stimulation
- Healthy children (4-11y) (Experimental)
  Interventions: Other: Down-phase targeted auditory stimulation
- Healthy teenagers (12-17y) (Experimental)
  Interventions: Other: Down-phase targeted auditory stimulation
- Healthy young adults (18-30y) (Experimental)
  Interventions: Other: Down-phase targeted auditory stimulation

INTERVENTIONS:
Other: Down-phase targeted auditory stimulation — The presentation of a soft, brief tone (50 ms of pink noise). The volume will be held low enough to avoid provoking arousals or awakenings. In case of a waking-up-reaction, the volume will be lowered in steps of 5 dB.

SUMMARY:
Sleep slow waves (SSW) and the pathophysiological mechanisms of spike generation in patients with epilepsy are tightly linked. SSW are cortically generated oscillations (~1 Hz) alternating between a hyperpolarized down-state (neuronal silence) and a depolarized up-state (neuronal firing). It has been shown experimentally that with increasing synchrony of slow neuronal oscillations, spike wave occurrence is facilitated. Auditory stimulation applied in correspondence to the SSW "up-phase" may increase the amplitude of the following SSW. Contrarywise, tones applied at the SSW "down-phase" may have a disruptive effect on SSW.

Participants: Patients with epilepsy with epileptic discharges in their sleep EEG, as well as healthy controls

Objective: Characterizing the effects of down-phase-targeted auditory stimulation on behavior and sleep EEG characteristics and determine whether the changes in sleep EEG characteristics are associated with the changes in behavior and wake EEG characteristics.

DETAILED DESCRIPTION:
The investigators aim to evaluate the effect of closed-loop auditory stimulation during sleep in healthy children, adolescents and adults, as well children, adolescents and adults with epilepsy. During closed-loop auditory stimulation, a brief, quiet, non-arousing auditory stimuli, e.g. brief bursts of pink noise (50ms), are presented at specific moments during sleep. This procedure allows to noninvasively interact with endogenous brain activity and to influence sleep-dependent neuroplasticity.

Sleep slow waves (SSW) and the pathophysiological mechanisms of spike generation in patients with epilepsy are tightly linked. SSW are cortically generated oscillations (~1 Hz) alternating between a hyperpolarized down-state (neuronal silence) and a depolarized up-state (neuronal firing). It has been shown experimentally that with increasing synchrony of slow neuronal oscillations, spike wave occurrence is facilitated. Auditory stimulation applied in correspondence to the SSW "up-phase" may increase the amplitude of the following SSW. Contrarywise, tones applied at the SSW "down-phase" may have a disruptive effect on SSW.

In a control week participants' usual sleeping behavior will be assessed using activity meters and sleep diaries. During the lab visits, sleep and wake brain activity will be measured using EEG at the sleep laboratory. For sleep recordings, other standard polysomnographic (PSG) measures will be recorded as well. Within the study, further measures include a structural MRI, IQ, as well as motor, cognitive, and vigilance tests. Participants' well-being and tolerance to the intervention will be assessed with questionnaires.

Thus, the investigators will have the following source data: PSG data, computer based test results (cognitive functioning, vigilance, memory and motor tests), IQ and questionnaire data, actigraphy data, and, depending on the participant and the availability of the MRI scanner, structural MRI data.

The sample size of the study is based on previous publications showing a significant effect of closed-loop auditory stimulation on NREM sleep EEG markers and declarative memory consolidation (Ngo et al., 2013). By including 11 participants they could demonstrate significant results both for the behavioral and electrophysiological data. Therefore, the investigators assume that it would be statistically meaningful to recruit at least 20 subjects per age group.

As the goal is to record 160 complete datasets, all these datasets will be used for the analysis. Incomplete datasets due to early withdrawal can be included partially for analyses in which only the available measures are included.

For any given analysis, datasets missing the relevant data will be excluded. The investigators will ensure that no analysis is based on less than 90% of the pursued sample size, meaning that at least 18 datasets per age and health group will enter all analyses (healthy participants or patients with epilepsy of a particular age group). In other words, no more than two participants would be excluded between outliers and missing data. Should this be exceeded, the investigators will compensate by recruiting additional participants

The data quality will be checked immediately after each experimental session to confirm the correct timing of presented sounds, as well as to assess the effect of closed-loop auditory stimulation on sleep EEG markers. The experiment will be continued if there will be a significant change in slow-wave activity in the first 10 participants (p < 0.05, paired-samples t-test) associated with closed-loop auditory stimulation application. The final analysis described in the section below will be performed after all the data is collected.

All study data will be archived at University Children's Hospital for a minimum of 10 years after study termination or premature termination of the clinical trial. The anonymized EEGs are stored on the server of the EEG division of the University Children's Hospital.

Data generation, transmission, archiving and analysis strictly follows the current Swiss legal requirements for data protection. Personal identifiable information will be handled with complete confidentiality and will only be accessible to authorized personnel who require such information to fulfill their duties within the scope of the research project. The documents of the telephone interview are kept enclosed. On the project specific documents, participants are only identified by a unique participant number. Participant IDs and corresponding names will be saved in an encrypted participant identification list, accessible only to the Principal Investigator and authorized members of the team.

The Sponsor-Investigator is implementing and maintaining quality assurance and quality control systems with written SOPs and Working Instructions to ensure that trials are conducted and data are generated, documented (record), and reported in compliance with the protocol, GCP, and applicable regulatory requirement(s). Monitoring and audits will be conducted during the course of the study for quality assurance purposes. The day-to-day management of the study will be coordinated through the selected PhD student supervised by the postdoctoral researcher.

The investigator will allow the persons being responsible for the audit or the inspection to have access to the source data/documents and to answer any questions arising. All involved parties will keep the patient data strictly confidential.

ELIGIBILITY:
Inclusion criteria

* Participants of any gender
* Children, adolescents and young adults (4-30 years old)
* Right-handed
* Written informed consent by the participant or, if applicable, by their legal guardian after receiving information about the study For healthy participants:
* Good general health status

For patients with epilepsy:

* Diagnosed with epilepsy
* Wake or sleep EEG within the last 12 months showing epileptic discharges.
* Attending a regular school.

Exclusion criteria

* Irregular sleep-wake rhythm
* Shift work
* Daytime sleep
* Excessive sweating
* Obesity
* Sleep, psychiatric, neurological or physical disorders or illnesses other than epilepsy
* Hearing disorder
* Travelling across 2 or more time zones within the last month
* Pregnancy
* Skin allergy or very sensitive skin
* Drug and medication use or abuse other than for the treatment of epilepsy
* Daily nicotine use
* High caffeine consumption, including coffee, black and green tea, mate, cola, energy drinks, and iced tea

  * <16 years: >1 servings/day = >80 mg caffeine
  * >=16 years: >2 servings/day = >160 mg caffeine
* Alcohol consumption

  * <16 years: any alcohol
  * 16-17 years: >3-4 standard servings per week
  * >=18 years: >1 standard serving per day (>14 mg)
* Inability to follow the procedures of the study For patients with epilepsy:
* Epilepsy syndromes with a high risk of seizure occurrence during the study night
* Generalized motor and/or focal motor seizure frequency >1/week
* Generalized motor and/or focal motor seizure within 24h before the study night
* History of convulsive status epilepticus
* History of seizures provoked by sleep deprivation
* Treatment with corticosteroids, immunosuppressants or vagus nerve stimulation

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CLAS on EEG characteristics & behavior | Up to 4 years
  CLAS changes sleep EEG characteristics (slow-wave and spindle activity) and the measured behavior (e.g. cognitive, memory and motor performance).
EEG characteristics on behavior & wake EEG characteristics | Up to 4 years
  The changes in sleep EEG characteristics (slow-wave and spindle activity) correlate with the changes in measured behavior (attention [TAP battery], reaction time [TAP battery], and declarative [word-pair memory task] & spatial memory [object-location task]) and wake EEG characteristics (frequencies up to 40 Hz).

SECONDARY OUTCOMES:
Performance in attention in epilepsy patients | Up to 4 years
  Attention (measured with TAP battery) of patients with epilepsy is restored to the level of healthy participants of the same age.
Performance in reaction times in epilepsy patients | Up to 4 years
  Reaction times (measured with TAP battery) of patients with epilepsy is restored to the level of healthy participants of the same age.
Performance in spatial memory in epilepsy patients | Up to 4 years
  Spatial memory (measured with object-location task) of patients with epilepsy is restored to the level of healthy participants of the same age.
Performance in declarative memory in epilepsy patients | Up to 4 years
  Declarative memory (measured with word-pair memory task) of patients with epilepsy is restored to the level of healthy participants of the same age.
CLAS on sleep slow waves | Up to 4 years
  Qualitative exploration of CLAS effect on the sleep slow waves across different age groups.
CLAS on other sleep EEG characteristics, such as sleep spindles | Up to 4 years
  Qualitative exploration of CLAS effect on other sleep EEG characteristics, such as sleep spindles across different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Huber, Prof. Dr., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Voluntary approval of the participant or legal guardian of the participant is given by signed informed consent. Personal data will be collected and immediately coded to provide strict confidentiality. The participant code will only be available to the principal investigator and research coordinators. The EEG data, completely anonymized, will be made publicly available to be used in other studies, for which the participant must provide separate consent. The investigators comply with all legal provisions of the Data Protection Act.
  The data, fully anonymized, will be published in a dedicated online repository. The data includes
  * PSG data + CLAS triggers
  * Basic demographic information: gender, age, socioeconomic status, handedness
  * Chronotype score
  * Responses to behavioral tests
  * Actigraphy
  * Sleep quality and sleepiness scores
Time Frame: Start: December 2019 End: December 2025
Access Criteria: Ideally, the investigators would like to publish the data through the University of Zurich, which is currently in the process of developing and contributing to the SWISSUbase. Unfortunately, at this time, the repository for neural, biological or psychology data has not yet been created. If, by the time of publication, this is still unavailable, the investigators will choose a repository that is compliant with the FAIR principles such as OpenNeuro. At the end of the project the investigators will evaluate the infrastructures available; it is conceivable that a Swiss university resource, or more suitable repository, will be established by then.
URL: https://info.swissubase.ch

REFERENCES:
- [Background] Bellesi M, Riedner BA, Garcia-Molina GN, Cirelli C, Tononi G. Enhancement of sleep slow waves: underlying mechanisms and practical consequences. Front Syst Neurosci. 2014 Oct 28;8:208. doi: 10.3389/fnsys.2014.00208. eCollection 2014. PMID 25389394
- [Background] Bolsterli BK, Gardella E, Pavlidis E, Wehrle FM, Tassinari CA, Huber R, Rubboli G. Remission of encephalopathy with status epilepticus (ESES) during sleep renormalizes regulation of slow wave sleep. Epilepsia. 2017 Nov;58(11):1892-1901. doi: 10.1111/epi.13910. Epub 2017 Sep 27. PMID 28960278
- [Background] Bolsterli BK, Schmitt B, Bast T, Critelli H, Heinzle J, Jenni OG, Huber R. Impaired slow wave sleep downscaling in encephalopathy with status epilepticus during sleep (ESES). Clin Neurophysiol. 2011 Sep;122(9):1779-87. doi: 10.1016/j.clinph.2011.01.053. Epub 2011 Mar 26. PMID 21441067
- [Background] Bolsterli Heinzle BK, Fattinger S, Kurth S, Lebourgeois MK, Ringli M, Bast T, Critelli H, Schmitt B, Huber R. Spike wave location and density disturb sleep slow waves in patients with CSWS (continuous spike waves during sleep). Epilepsia. 2014 Apr;55(4):584-91. doi: 10.1111/epi.12576. Epub 2014 Mar 20. PMID 24650120
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Esser SK, Hill SL, Tononi G. Sleep homeostasis and cortical synchronization: I. Modeling the effects of synaptic strength on sleep slow waves. Sleep. 2007 Dec;30(12):1617-30. doi: 10.1093/sleep/30.12.1617. PMID 18246972
- [Background] Fattinger S, de Beukelaar TT, Ruddy KL, Volk C, Heyse NC, Herbst JA, Hahnloser RHR, Wenderoth N, Huber R. Deep sleep maintains learning efficiency of the human brain. Nat Commun. 2017 May 22;8:15405. doi: 10.1038/ncomms15405. PMID 28530229
- [Background] Fattinger S, Heinzle BB, Ramantani G, Abela L, Schmitt B, Huber R. Closed-Loop Acoustic Stimulation During Sleep in Children With Epilepsy: A Hypothesis-Driven Novel Approach to Interact With Spike-Wave Activity and Pilot Data Assessing Feasibility. Front Hum Neurosci. 2019 May 21;13:166. doi: 10.3389/fnhum.2019.00166. eCollection 2019. PMID 31164813
- [Background] Fattinger S, Schmitt B, Bolsterli Heinzle BK, Critelli H, Jenni OG, Huber R. Impaired slow wave sleep downscaling in patients with infantile spasms. Eur J Paediatr Neurol. 2015 Mar;19(2):134-42. doi: 10.1016/j.ejpn.2014.11.002. Epub 2014 Nov 29. PMID 25530030
- [Background] Frauscher B, von Ellenrieder N, Ferrari-Marinho T, Avoli M, Dubeau F, Gotman J. Facilitation of epileptic activity during sleep is mediated by high amplitude slow waves. Brain. 2015 Jun;138(Pt 6):1629-41. doi: 10.1093/brain/awv073. Epub 2015 Mar 19. PMID 25792528
- [Background] Galer S, Urbain C, De Tiege X, Emeriau M, Leproult R, Deliens G, Nonclerq A, Peigneux P, Van Bogaert P. Impaired sleep-related consolidation of declarative memories in idiopathic focal epilepsies of childhood. Epilepsy Behav. 2015 Feb;43:16-23. doi: 10.1016/j.yebeh.2014.11.032. Epub 2014 Dec 26. PMID 25546732
- [Background] Halasz P, Bodizs R, Ujma PP, Fabo D, Szucs A. Strong relationship between NREM sleep, epilepsy and plastic functions - A conceptual review on the neurophysiology background. Epilepsy Res. 2019 Feb;150:95-105. doi: 10.1016/j.eplepsyres.2018.11.008. Epub 2019 Jan 31. PMID 30712997
- [Background] Huber R, Ghilardi MF, Massimini M, Tononi G. Local sleep and learning. Nature. 2004 Jul 1;430(6995):78-81. doi: 10.1038/nature02663. Epub 2004 Jun 6. PMID 15184907
- [Background] Ngo HV, Martinetz T, Born J, Molle M. Auditory closed-loop stimulation of the sleep slow oscillation enhances memory. Neuron. 2013 May 8;78(3):545-53. doi: 10.1016/j.neuron.2013.03.006. Epub 2013 Apr 11. PMID 23583623
- [Background] Vyazovskiy VV, Harris KD. Sleep and the single neuron: the role of global slow oscillations in individual cell rest. Nat Rev Neurosci. 2013 Jun;14(6):443-51. doi: 10.1038/nrn3494. Epub 2013 May 2. PMID 23635871
- [Background] Vyazovskiy VV, Olcese U, Lazimy YM, Faraguna U, Esser SK, Williams JC, Cirelli C, Tononi G. Cortical firing and sleep homeostasis. Neuron. 2009 Sep 24;63(6):865-78. doi: 10.1016/j.neuron.2009.08.024. PMID 19778514
- Available data/document: Individual Participant Data Set — https://info.swissubase.ch